CLINICAL TRIAL: NCT05913206
Title: Developing an Innovative Decision Support Tool for Pediatric Neuromuscular Scoliosis- Aim 1
Brief Title: Understanding Factors in Decision Making for Children with Medical Complexity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Utah (Other)
Collaborators: Children's Hospital Los Angeles (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Health Services Research
Other Study IDs: 00154724
Record Dates: First submitted 2023-06-12; First posted 2023-06-22 (Actual); Last update posted 2024-10-18 (Actual); Status verified 2023-10

CONDITIONS: Multiple Chronic Conditions; Children with Medical Complexity
Keywords: Shared decision making; Health communication; Patient- and Family-Centered Care
MeSH Terms: conditions — Multiple Chronic Conditions | interventions — Narrative Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Participants and the investigator team will be blinded to which condition the participant is randomized.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (16):
- Control (No Intervention): No new communication approaches received.
- Ambiguity only (Experimental): Receive information about ambiguity related to the clinical decision.
  Interventions: Behavioral: Ambiguity
- Ambiguity and complexity only (Experimental): Receive information about ambiguity and complexity related to the clinical decision.
  Interventions: Behavioral: Ambiguity; Behavioral: Complexity
- Ambiguity and normalizing only (Experimental): Receive information about ambiguity and normalizing language related to the clinical decision.
  Interventions: Behavioral: Ambiguity; Behavioral: Normalizing language
- Ambiguity, complexity, and normalizing only (Experimental): Receive information about ambiguity, complexity, and normalizing language related to the clinical decision.
  Interventions: Behavioral: Ambiguity; Behavioral: Complexity; Behavioral: Normalizing language
- Complexity only (Experimental): Receive information about complexity related to the clinical decision.
  Interventions: Behavioral: Complexity
- Complexity and normalizing only (Experimental): Receive information about complexity and normalizing language related to the clinical decision.
  Interventions: Behavioral: Complexity; Behavioral: Normalizing language
- Normalizing only (Experimental): Receive information about normalizing language related to the clinical decision.
  Interventions: Behavioral: Normalizing language
- Narratives only (Experimental): Receive narratives in addition to the control condition.
  Interventions: Behavioral: Narrative
- Ambiguity and narratives only (Experimental): Receive information about ambiguity and narratives related to the clinical decision.
  Interventions: Behavioral: Ambiguity; Behavioral: Narrative
- Ambiguity, complexity, and narratives only (Experimental): Receive information about ambiguity, complexity, and narratives related to the clinical decision.
  Interventions: Behavioral: Ambiguity; Behavioral: Complexity; Behavioral: Narrative
- Ambiguity, normalizing, and narratives only (Experimental): Receive information about ambiguity, normalizing language, and narratives related to the clinical decision.
  Interventions: Behavioral: Ambiguity; Behavioral: Normalizing language; Behavioral: Narrative
- All (Experimental): Receive all new communication approaches
  Interventions: Behavioral: Ambiguity; Behavioral: Complexity; Behavioral: Normalizing language; Behavioral: Narrative
- Complexity and narratives only (Experimental): Receive information about complexity and narratives related to the clinical decision.
  Interventions: Behavioral: Complexity; Behavioral: Narrative
- Complexity, normalizing, and narratives only (Experimental): Receive information about complexity, normalizing language, and narratives related to the clinical decision.
  Interventions: Behavioral: Complexity; Behavioral: Normalizing language; Behavioral: Narrative
- Normalizing and narratives only (Experimental): Receive information about normalizing language and narratives related to the clinical decision.
  Interventions: Behavioral: Normalizing language; Behavioral: Narrative

INTERVENTIONS:
Behavioral: Ambiguity — The intervention is a novel communication approach to communicate ambiguity related to the potential risks and benefits associated with clinical decision making for parents and caregivers of children with medical complexity.
  Arms: All; Ambiguity and complexity only; Ambiguity and narratives only; Ambiguity and normalizing only; Ambiguity only; Ambiguity, complexity, and narratives only; Ambiguity, complexity, and normalizing only; Ambiguity, normalizing, and narratives only
Behavioral: Complexity — The intervention is a novel communication approach to communicate complexity related to the potential risks and benefits associated with clinical decision making for parents and caregivers of children with medical complexity.
  Arms: All; Ambiguity and complexity only; Ambiguity, complexity, and narratives only; Ambiguity, complexity, and normalizing only; Complexity and narratives only; Complexity and normalizing only; Complexity only; Complexity, normalizing, and narratives only
Behavioral: Normalizing language — The intervention is a novel communication approach to normalize and explain the inherent uncertainty faced by parents of children with medical complexity during clinical decision making.
  Arms: All; Ambiguity and normalizing only; Ambiguity, complexity, and normalizing only; Ambiguity, normalizing, and narratives only; Complexity and normalizing only; Complexity, normalizing, and narratives only; Normalizing and narratives only; Normalizing only
Behavioral: Narrative — Parent and caregiver narratives about their decision making experiences for the care of their child with medical complexity.
  Arms: All; Ambiguity and narratives only; Ambiguity, complexity, and narratives only; Ambiguity, normalizing, and narratives only; Complexity and narratives only; Complexity, normalizing, and narratives only; Narratives only; Normalizing and narratives only

SUMMARY:
The goal of this clinical trial is to compare different strategies to communicate around potential risks and benefits related to treatment decision making in parents/adult caregivers of children with medical complexity. The objective of this study is to identify the most effective ways to communicate decision-related risks and benefits to improve the quality of caregiver decision making for children with medical complexity.

Participants will view a video of a simulated clinic visit and related medical information and complete a survey about their experiences. Researchers will compare participant survey responses to see if decision quality changes based on the information reviewed by the participant.

DETAILED DESCRIPTION:
Children with medical complexity, their caregivers, and their providers face a multitude of complex, high stakes medical decisions throughout their lifetime. Best practices for the provision of high quality shared decision making in the care of children with medical complexity do not exist. Unique challenges to support decision making for caregivers of children with medical complexity include communication of decision-related risks and benefits and knowledge related to the decision. This study will test the efficacy of various communication techniques in the setting of a simulated patient encounter.

ELIGIBILITY:
Inclusion Criteria:

* Adult caregiver of a child with medical complexity
* English- or Spanish-speaking

Exclusion Criteria:

* Child is diagnosed with neuromuscular scoliosis but has not yet made a decision about whether to undergo spinal fusion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 826 (Actual)
Dates: Start 2023-06-29 (Actual); Primary Completion 2024-08-29 (Actual); Study Completion 2024-08-29 (Actual)

PRIMARY OUTCOMES:
Decision readiness | Immediately after reviewing the intervention
  Differences in decision readiness between arms as measured by the validated PrepDM survey measure. The PrepDM is a 10-item (1 to 5 scale) validated survey measure that evaluates a patient's perceived readiness to make a decision with their healthcare provider. The composite score is a mean of all items converted to a scale of 0-100 with higher scores indicating greater decision readiness. PrepDM is widely used to evaluate the effectiveness of decision aids.

SECONDARY OUTCOMES:
Decisional Conflict Scale | Immediately after reviewing the intervention
  Difference in decisional conflict score between arms. The decisional conflict scale is a 16-item (1-5 scale) validated survey measure that evaluates a participant's decisional conflict about a decision that is made and includes five subdomains (uncertainty, informed, values clarity, support, and effective decision). Total and subdomain scores are calculated using a mean composite score and transformed to a scale of 0 to 100 with higher scores indicating higher decisional conflict.
Decision intent for treatment | Immediately after reviewing the intervention
  Proportion of participants selecting surgery between the arms.
Knowledge | Immediately after reviewing the intervention
  Difference in mean score of total knowledge questions answered correctly between arms. The score will be calculated from 5 knowledge questions.

CONTACTS AND LOCATIONS:
Overall Officials: Jody L Lin, MD, MS, Principal Investigator — University of Utah
Locations (2):
- United States (2):
  - Children's Hospital Los Angeles, Los Angeles, California
  - University of Utah, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No